CLINICAL TRIAL: NCT06789770
Title: The Impact of Nasal Versus Oral Breathing on Measures of Drug-Induced Sleep Endoscopy
Brief Title: Nasal vs Oral Breathing in Drug Induced Sleep vs Natural Sleep
Acronym: Nasal vs Oral
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: McCabe Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: 857046
Record Dates: First submitted 2024-11-13; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: breathing route; OSA; nasal breathing; oral breathing
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will provide important new information regarding (1) the relationship between route of breathing and airway collapsibility and (2) whether route of breathing during DISE (Drug-Induced Sleep Endoscopy) is representative of natural sleep.

DETAILED DESCRIPTION:
As part of standard of care, a drug-induced sleep endoscopy will be done, where route of breathing will be determined as a percentage of total breaths (during baseline, lateral sleep and maneuver). As part of the research procedure, an in-laboratory Polysomnogram will be conducted as study procedure including a oronasal pressure signal cannula to assess route of breathing.

ELIGIBILITY:
Inclusion Criteria:

* • Adults (≥ 18yrs) that underwent clinical evaluation at the CPAP Alternatives Clinic at Penn Otorhinolaryngology.

  * Must have at least mild OSA (AHI>5)

Exclusion Criteria:

* • Sleep study with an AHI<5, >25% of total events being central or mixed events, or inability to achieve adequate drug-induced sleep.

  * Upper Respiratory Illness at the time of the DISE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are referred to the PI's CPAP alternatives clinic. They are of all ages (18+) and all genders.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Is someone a mouth or nose breather? What kind of airway obstruction and collapse do they have? | During the DISE (30 minutes)
  Naming where the sites of obstruction are during DISE (by collecting a VOTE score) and noting whether the route of breathing is oral or nasal.

SECONDARY OUTCOMES:
Is a patients route of breathing the same during DISE and PSG? | During DISE (30 minutes) and PSG (1 night sleep study)
  Compare route of breathing (oral, nasal or mixed) in DISE or in PSG.

CONTACTS AND LOCATIONS:
Overall Officials: Julianna Rodin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided